CLINICAL TRIAL: NCT02852876
Title: A Double-Blind, Placebo-Controlled Single Dose Escalating Study to Assess the Safety, Tolerability and Pharmacokinetics of ASP2151 in Healthy Male Subjects, Followed by an Open, Two-Period Crossover Study to Assess the Effect of Fed Conditions on the Safety, Tolerability and Pharmacokinetics of ASP2151
Brief Title: Study to Evaluate the Safety and Pharmacokinetics of Single Doses of ASP2151 in Healthy Male Subjects and the Effects of Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 15L-CL-002; 2005-002697-30 (EudraCT Number)
Record Dates: First submitted 2016-07-29; First posted 2016-08-02 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Herpes Genitalis; Herpes Zoster
Keywords: Safety of ASP2151; Phase 1; Pharmacokinetics; Healthy male subjects; Tolerability; Food effect of ASP2151
MeSH Terms: conditions — Herpes Genitalis; Herpes Zoster | interventions — ASP2151

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (11):
- Part 1: ASP2151 Single Ascending Dose Group A (Fasting) (Experimental): Participants will receive single dose of ASP2151 assigned to Group A on day 1
  Interventions: Drug: ASP2151
- Part 1: ASP2151 Single Ascending Dose Group B (Fasting) (Experimental): Participants will receive single dose of ASP2151 assigned to Group B on day 1
  Interventions: Drug: ASP2151
- Part 1: ASP2151 Single Ascending Dose Group C (Fasting) (Experimental): Participants will receive single dose of ASP2151 assigned to Group C on day 1
  Interventions: Drug: ASP2151
- Part 1: ASP2151 Single Ascending Dose Group D (Fasting) (Experimental): Participants will receive single dose of ASP2151 assigned to Group D on day 1
  Interventions: Drug: ASP2151
- Part 1: ASP2151 Single Ascending Dose Group E (Fasting) (Experimental): Participants will receive single dose of ASP2151 assigned to Group E on day 1
  Interventions: Drug: ASP2151
- Part 1: ASP2151 Single Ascending Dose Group F (Fasting) (Experimental): Participants will receive single dose of ASP2151 assigned to Group F on day 1
  Interventions: Drug: ASP2151
- Part 1: Placebo Single Ascending Dose (Fasting) (Placebo Comparator): Participants will receive single dose of matching placebo on day 1
  Interventions: Drug: Placebo
- Part 2: ASP2151 (Fasting) (Experimental): Participants will receive a single dose of ASP2151 under fasted conditions on day 1 in the first treatment period (period 1). Following a wash-out period of at least five days, the treatment will be repeated in the reverse orientation (period 2)
  Interventions: Drug: ASP2151
- Part 2: ASP2151 (Fed) (Experimental): Participants will receive a single dose of ASP2151 under fed conditions on day 1 in the first treatment period (period 1). Following a wash-out period of at least five days, the treatment will be repeated in the reverse orientation (period 2)
  Interventions: Drug: ASP2151
- Part 1: ASP2151 Single Ascending Dose Group G (Fasting) (Experimental): Participants will receive single dose of ASP2151 assigned to Group G on day 1
  Interventions: Drug: ASP2151
- Part 1: ASP2151 Single Ascending Dose Group H (Fasting) (Experimental): Participants will receive single dose of ASP2151 assigned to Group H on day 1
  Interventions: Drug: ASP2151

INTERVENTIONS:
Drug: ASP2151 — Oral
  Arms: Part 1: ASP2151 Single Ascending Dose Group A (Fasting); Part 1: ASP2151 Single Ascending Dose Group B (Fasting); Part 1: ASP2151 Single Ascending Dose Group C (Fasting); Part 1: ASP2151 Single Ascending Dose Group D (Fasting); Part 1: ASP2151 Single Ascending Dose Group E (Fasting); Part 1: ASP2151 Single Ascending Dose Group F (Fasting); Part 1: ASP2151 Single Ascending Dose Group G (Fasting); Part 1: ASP2151 Single Ascending Dose Group H (Fasting); Part 2: ASP2151 (Fasting); Part 2: ASP2151 (Fed)
Drug: Placebo — Oral
  Arms: Part 1: Placebo Single Ascending Dose (Fasting)

SUMMARY:
The objective of this study is to evaluate the safety and tolerability of single rising doses of ASP2151 under fasted condition in healthy male subjects.

The study will also evaluate the pharmacokinetics (PK) of a single dose of ASP2151 under fasted versus fed conditions in healthy male subjects.

DETAILED DESCRIPTION:
Study will be divided into two parts. Part 1 will evaluate the safety and tolerability of ASP2151 single rising doses in groups A-H in fasted condition and to determine the maximum tolerable dose (MTD) if possible.

Part 2 will evaluate the effect of fasted versus fed conditions on the safety, tolerability and PK of a single dose of ASP2151 in two treatment cycles. The wash-out period between the two treatment cycles will be at least 5 days and not shorter than five times the average elimination half-life of ASP2151, as determined in part 1 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Body weight between 60 and 100 kg, and BMI between 18 and 30 kg/m2 inclusive

Exclusion Criteria:

* Known or suspected hypersensitivity to ASP2151 or any components of the formulation used
* Any clinically significant history of asthma, eczema, any other allergic condition or previous severe hypersensitivity to any drug
* Any clinically significant history of genital herpes symptoms and/or herpes zoster symptoms in the 3 months prior to admission to the Clinical Unit
* Any clinically significant history of any other disease or disorder - gastrointestinal, cardiovascular, respiratory, renal, hepatic, neurological, dermatological, psychiatric or metabolic
* Abnormal pulse rate and/or blood pressure measurements at the pre-study visit as follows: Pulse rate <40 or >90 bpm (beats per minute); mean systolic blood pressure <90 or >140 mmHg (millimeter of mercury); mean diastolic blood pressure <40 or >95 mmHg
* Regular use of any prescribed or OTC (over the counter) drugs in the 4 weeks prior to admission to the Clinical Unit OR any use of such drugs in the 2 weeks prior to admission to the Clinical Unit
* Any use of drugs of abuse within 3 months prior to admission to the Clinical Unit
* History of smoking more than 10 cigarettes per day within 3 months prior to admission to the Clinical Unit
* History of drinking more than 21 units of alcohol per week within 3 months prior to admission to the Clinical Unit
* Donation of blood or blood products within 3 months, prior to admission to the Clinical Unit
* Positive serology test for HBsAg (Hepatitis B surface antigen), HAV IgM (Hepatitis A Virus), anti-HCV (Hepatitis C Virus) or anti-HIV (Human Immunodeficiency Virus) 1 and 2
* Not willing or able to swallow size 00 capsules

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2005-09; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed by nature, frequency, and severity of Adverse Events (AEs) | Up to Day 15 of each treatment period
  For Part 1 and Part 2
Safety assessed by 12- lead electrocardiogram (ECG) | Up to Day 15 of each treatment period
  For Part 1 and Part 2
Safety assessed by vital sign measurement: blood pressure | Up to Day 15 of each treatment period
  For Part 1 and Part 2 includes systolic and blood diastolic pressure
Safety assessed by vital sign measurement: pulse rate | Up to Day 15 of each treatment period
  For Part 1 and Part 2
Safety assessed by laboratory test: biochemical | Up to Day 15 of each treatment period
  For Part 1 and Part 2
Safety assessed by laboratory test: hematological | Up to Day 15 of each treatment period
  For Part 1 and Part 2
Safety assessed by laboratory test: serology | Up to Day 15 of each treatment period
  For Part 1 and Part 2
Safety assessed by laboratory test: urinalysis | Up to Day 15 of each treatment period
  For Part 1 and Part 2
Safety assessed by physical exam: body weight | Up to Day 15 of each treatment period
  For Part 1 and Part 2
Safety assessed by physical exam: height | Up to Day 15 of each treatment period
  For Part 1 and Part 2
Safety assessed by physical exam: body mass index (BMI) | Up to Day 15 of each treatment period
  For Part 1 and Part 2

SECONDARY OUTCOMES:
Pharmacokinetics of ASP2151 in plasma: AUC0-inf | Up to 48 hours in each treatment period
  For Part 1 and 2. AUC0-inf: Area under the concentration time curve from the time of dosing extrapolated to time infinity
Pharmacokinetics of ASP2151 in plasma: t1/2 | Up to 48 hours in each treatment period
  For Part 1 and 2. t1/2: Apparent terminal elimination half-life
Pharmacokinetics of ASP2151 in plasma: Cmax | Up to 48 hours in each treatment period
  For Part 1 and 2. Cmax: Maximum concentration
Pharmacokinetics of ASP2151 in plasma: tmax | Up to 48 hours in each treatment period
  For Part 1 and 2. tmax: The time after dosing when Cmax occurs
Pharmacokinetics of ASP2151 in plasma: CL/F | Up to 48 hours in each treatment period
  For Part 1 and 2. CL/F: Oral clearance
Pharmacokinetics of ASP2151 in plasma: Vz/F | Up to 48 hours in each treatment period
  For Part 1 and 2. Vz/F: Apparent volume of distribution
Pharmacokinetics of ASP2151 in plasma: AUClast | Up to 48 hours in each treatment period
  For Part 1 and 2. AUClast: Area under the plasma concentration time curve from time of dosing up to the last quantifiable sample
Pharmacokinetics of ASP2151 in plasma: tlag | Up to 48 hours in each treatment period
  For Part 1 and 2. tlag: Absorption lag time
Pharmacokinetics of ASP2151 in urine: Aelast | Up to 48 hours in each treatment period
  For Part 1 and 2. Aelast: Amount excreted unchanged in urine from time of dosing up to the last quantifiable sample
Pharmacokinetics of ASP2151 in urine: Ae0-inf | Up to 48 hours in each treatment period
  For Part 1 and 2. Ae0-inf: Amount excreted unchanged in urine from time of dosing extrapolated to infinity
Pharmacokinetics of ASP2151 in urine: Ae% | Up to 48 hours in each treatment period
  For Part 1 and 2. Ae%: Percent of ASP2151 amount excreted in urine
Pharmacokinetics of ASP2151 in urine: CLr | Up to 48 hours in each treatment period
  For Part 1 and 2. CLr: Renal clearance

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Clinical Pharmacology & Exploratory Dev.
Locations (1):
- Site FR1717, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kusawake T, Keirns JJ, Kowalski D, den Adel M, Groenendaal-van de Meent D, Takada A, Ohtsu Y, Katashima M. Pharmacokinetics and Safety of Amenamevir in Healthy Subjects: Analysis of Four Randomized Phase 1 Studies. Adv Ther. 2017 Dec;34(12):2625-2637. doi: 10.1007/s12325-017-0642-4. Epub 2017 Nov 13. PMID 29134426